CLINICAL TRIAL: NCT06972199
Title: The Effect of Reflexology Massage and Hot Water Foot Bath on Pain and Gastrointestinal Functions After Colorectal Surgery
Brief Title: Reflexology Massage and Hot Water Foot Bath for Pain and GI Recovery After Colorectal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Cansu Mert, Doctoral Student, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18.2024fbu
Record Dates: First submitted 2025-04-29; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Surgery; Reflexology; Traditional Chinese Medication (TCM); Nursing
MeSH Terms: interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reflexology (Experimental): Reflexology application
  Interventions: Behavioral: Reflexology
- Hot water foot bath (Experimental): Hot water foot bath application
  Interventions: Behavioral: Hot water foot bath
- Control (No Intervention): There will be no intervention

INTERVENTIONS:
Behavioral: Reflexology — Reflexology application
  Arms: Reflexology
Behavioral: Hot water foot bath — Hot water foot bath application
  Arms: Hot water foot bath

SUMMARY:
This study was planned to examine the effect of non-invasive treatment methods that can be applied to alleviate complications involving gastrointestinal system functions such as pain, nausea, vomiting, and absence of gas/faecal output after colorectal (colon and rectum) cancer surgery. The two main intervention methods of the study were reflexology massage and hot water foot bath. The effects of these methods on reducing postoperative pain and improving gastrointestinal functions will be investigated. The study was planned as a randomised controlled experimental study to determine the effects of reflexology massage and hot water foot bath on postoperative pain and gastrointestinal functions in colorectal cancer patients undergoing laparoscopic surgery. It is thought that the study will provide evidence for determining the appropriate method to reduce pain and improve gastrointestinal functions in patients undergoing colorectal cancer surgery. The population of the study will consist of colorectal cancer patients who will undergo laparoscopic surgical intervention who are admitted to the General Surgery Clinic of SBU Istanbul Ümraniye Training and Research Hospital.

Based on the percentage measurement values of the methods to be studied in the literature review, G-POWER programme was used for sample calculation with an effect size of 0.4 (Cohen), 95% power and 0.05% margin of error. Cohen's standard effect size was taken as the basis for the effect size. The calculated value is the total value for 3 groups and the total sample size for 3 groups was found as n=102. The number of samples per group was determined as (n)=34. In order to prevent bias in the study, patients who meet the study criteria will be distributed to the experimental and control groups by computerised randomisation programme. Data will be collected by using the Patient Information Form consisting of two parts, Rhodes Nausea, Vomiting and Retching Index and Numerical Proportioning Scale (NRS) developed by the researcher in line with the literature. The data obtained will be evaluated with appropriate statistical methods in the licensed SPSS 21.0 package programme.

DETAILED DESCRIPTION:
This randomized controlled trial aims to evaluate the effectiveness of two non-pharmacological interventions-reflexology massage and hot water foot bath-on postoperative pain and gastrointestinal function in patients undergoing laparoscopic colorectal cancer surgery. The interventions will be applied in three groups: reflexology massage, hot water foot bath, and control group. Participants will be randomly assigned to groups using a computerized randomization method. Pain will be assessed using the Numerical Rating Scale (NRS), and gastrointestinal function will be evaluated through time to first gas and feces passage, as well as bowel sounds. Additionally, the Rhodes Index of Nausea, Vomiting, and Retching (RINVR) will be used to monitor symptoms related to postoperative nausea and vomiting. Data will also be collected using a researcher-developed Data Collection Form consisting of:

* Sociodemographic characteristics
* Medical and surgical history
* Postoperative vital signs (blood pressure, pulse, temperature, etc.)
* Gastrointestinal follow-up (bowel sounds per minute, time of first gas and feces output) This form was developed based on current literature and clinical practice guidelines and piloted prior to study launch. All data will be analyzed using SPSS 21.0.

The sample size was calculated using G*Power based on an effect size of 0.4 (Cohen), 95% power, and a 0.05 margin of error, resulting in 102 total participants (n=34 per group).

Ethical approval was obtained from the Non-Interventional Clinical Research Ethics Committee of Fenerbahçe University. The study is being conducted at the General Surgery Clinic of SBÜ Ümraniye Training and Research Hospital.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* Planning laparoscopic surgery for a malignant tumour in the large intestine,
* The same method was used for preoperative bowel and GI tract preparation,
* Postoperative Numerical Proportioning Scale (NRS) score of 3 and above,
* Verbal and written acceptance to participate in the research.

Exclusion Criteria:

* The patient has a temporary or permanent stoma,
* Having a history of reflexology application before,
* Open wound, infection, circulatory disorder, lesion, etc. in the areas where reflexology massage or hot water foot bath will be applied,
* Patient-controlled analgesia in the early postoperative period
* Having any problem that prevents verbal communication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain level | Within 24 hours postoperatively
  Postoperative pain levels of the participants will be measured with the Numerical Rating Scale (NRS), which ranges from 0 to 10, where 0 indicates no pain and 10 indicates the worst possible pain.
Gas release time | Within 24 hours postoperatively
  Time to first gas release of participants in the postoperative period after surgery

SECONDARY OUTCOMES:
Neusea | Within 24 hours postoperatively
  In the postoperative period, nausea and vomiting will be evaluated with the Rhodes Nausea, Vomiting and Retching Index (RNVRI), which has a total score range from 0 to 32. Higher scores indicate more severe symptoms.
Number of vomiting | Within 24 hours postoperatively
  The number of vomits occurring in the participants in the postoperative period will be recorded.

OTHER OUTCOMES:
Time to First Flatus | Within 48 hours postoperatively
  The time (in hours) from the end of surgery until the first passage of flatus, as recorded by the participant and verified by nursing staff. This value will be recorded in the Postoperative Bowel Function Monitoring Form.
Time to First Defecation | Within 72 hours postoperatively
  The time (in hours) from the end of surgery until the first defecation (bowel movement). Patients will self-report and nurses will document the exact time. Recorded in the postoperative bowel function table.
Time to Tolerate Oral Diet | within 24 hours postoperatively
  The time (in hours) from the end of surgery until the patient tolerates the first full oral diet without nausea or vomiting. Evaluated via dietary intake and nurse monitoring records.

CONTACTS AND LOCATIONS:
Overall Officials: Cansu Mert, Master, Principal Investigator — Istanbul University - Cerrahpasa
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul University-Cerrahpaşa, Istanbul, Istanbul
  - University of Health Sciences, Umraniye Training and Research Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: No